CLINICAL TRIAL: NCT05093140
Title: Anti-PD-1 Antibody (Camrelizumab) Plus R-CHOP Regimen for the Primary Extranodal Treatment-Naive Diffuse Large B Cell Lymphoma (CREDIT): a Prospective, Multicenter, Single-Arm, Phase II Trial
Brief Title: Camrelizumab Plus R-CHOP Regimen in Untreated Primary Extranodal DLBCL
Acronym: CREDIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-DLBCL-Ⅱ-004
Record Dates: First submitted 2021-10-11; First posted 2021-10-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Primary Extranodal Lymphoma; DLBCL
Keywords: primary extranodal lymphoma; DLBCL; R-CHOP; PD-1; camrelizumab
MeSH Terms: interventions — camrelizumab; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab+R-CHOP (Experimental): Induction therapy: camrelizumab in combination with rituximab Immunochemotherapy: rituximab, cyclophosphamide, hydroxyldaunorubicin, vincristine, prednisone Maintenance therapy: camrelizumab in patients achieved CR after immunotherapy
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Induction therapy:
  Camrelizumab 200mg, ivd, D1, Rituximab 375mg/m2, ivd, D1 every 3 weeks up to 2 cycles
  Immunochemotherapy:
  Rituximab: 375mg/m2, ivd, D1; Cyclophosphamide: 750mg/m2, iv or ivd, D1; Hydroxyldaunorubicin: 50mg/m2, iv or ivd, D1; Vincristine: 1.4 mg/m2 , iv(max：2mg), D1; Prednisone: 60mg/m2, po, d1-5 every 3 weeks up to 6 cycles Maintenance therapy: Camrelizumab 200mg, ivd, D1 every 4 weeks up to 6 cycles
  Other Names: Rituximab; Cyclophosphamide; Hydroxyldaunorubicin; Vincristine; Prednisone

SUMMARY:
To assess the efficacy and safety of camrelizumab combined with rituximab, vincristine, doxorubicin, cyclophosphamide and prednisone in the treatment of untreated primary extranodal DLBCL

ELIGIBILITY:
Inclusion Criteria:

* • Male or female patients: 18-65 years old.

  * Newly diagnosed patients
  * Primary extranodal lymphoma, histologically-confirmed DLBCL( including but not limited to follicular lymphoma grade 3B, or transformed DLBCL, EBV(+) DLBCL, ALK(+) DLBCL, high grade lymphoma). The primary site is limited to the gastrointestinal tract, nasal cavity and breast, and central nervous system( CNS) involvement must be excluded. Gastrointestinal tract involvement of DLBCL can be included in the group after evaluation without bleeding or perforation risk.
  * ECOG physical condition score: 0-2 points for patients.
  * The patients must be with at least one evaluable or measurable lesion meeting Lugano 2014 criteria, the evaluable lesion was: 18F fluorodeoxyglucose / positron emission tomography (18FDG-PET) examination showed that the uptake of extranodal areas was increased (higher than that of liver) and pet and / or computed. The features of tomography (CT) were in accordance with lymphoma. The measurable lesions were nodal lesions with a length of > 15 mm or extranodal lesions with a length of > 10 mm, accompanied by an increase in 18-FDG uptake. It is necessary to exclude the case where there is no measurable lesion and the diffuse 18-FDG uptake increase in the liver.
  * Hematology values must be within the following limits at baseline:

    1. Absolute neutrophil count (ANC) ≥1,500 cells/μL. In case bone marrow involvement, ANC≥1,000 cells/μL.
    2. Platelets≥75,000 cells/μL. In case bone marrow involvement, platelets≥50,000 cells/μL
    3. Hemoglobin≥90 g/L
  * Biochemical values must be within the following limits at baseline:

    1. Alanine aminotransferase（ALT）≤3×upper limit of normal (ULN).
    2. Aspartate aminotransferase (AST) ≤3×ULN
    3. Total bilirubin≤1.5×ULN, unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
    4. Serum creatinine ≤2×ULN or estimated Glomerular Filtration Rate ≥40/mL/min/1.73m2
  * LVEF within institutional normal limits, as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan.
  * Each subject (or their legally acceptable representative) must sigh an informed consent form (ICF) indicating that he or she understands the purpose of any procedures for the study and are willing to participate in the study.
  * Women of childbearing potential ( WOCBP) must have a negative serum (beta-human chorionic gonadotropin[β-hCG] ) or urine pregnancy test within 7 days before the first medication
  * Women of childbearing potential or men and their WOCBP partners should agree to take effective contraceptive measures from signing the ICF to 6 months after the last dose of study medication.

Exclusion Criteria:

- • Primary DLBCL arise in lymph nodes or other lymphatic tissues.

* Primary central nervous system lymphoma or secondary central nervous system involvement, known primary mediastinal lymphoma.
* A history of severe allergies or allergic reactions to humanized or murine monoclonal antibodies.
* In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known
* Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 1000 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 1000 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group.
* Patients with any active infections requiring systemic anti-infective treatment within 14 days of treatment.
* Received systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc..
* Received major surgery within 28 days before treatment or radiotherapy within 90 days before treatment.
* Received live vaccination (except influenza attenuated vaccine) within 28 days before treatment.
* Patients requiring long-term systemic glucocorticoid therapy or other immunosuppressive therapy (>prednisone 10mg/qd or equivalent dose of other glucocorticoid therapy). Allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy.
* Patients suffering from uncontrollable comorbid diseases, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or bleeding disorders.
* Pregnant or lactating women.
* Patients with a history of interstitial lung disease or non-infectious pneumonia. Subjects who have previously had drug-induced or radioactive non-infectious pneumonia but asymptomatic are allowed to enroll.
* Any life-threatening disease, physical condition or organ dysfunction according to the researchers' judgment may endanger the safety of the subject or put the clinical research at excessive risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 24 weeks

SECONDARY OUTCOMES:
Objective remission rate | six weeks
Objective remission rate | 24 weeks
Duration of Response | 2 years
  The time from the first assessment of CR or PR to PD (progressive disease) or death from any cause
Progression-free Survival | 2 years
  PFS was defined as time from study registration to first disease progression or death whichever occurred first, otherwise subject data were censored at time last known disease free
Overall Survival | 2 years
  OS was defined as time from study registration to death, and otherwise censored at time last known alive
Percentage of Participants With Adverse Events (AEs) | Up to 30 days after the last cycle of per-protocol treatment and 90 days after last dose of anti-PD-1 antibody
  Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, professor, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No